CLINICAL TRIAL: NCT03721640
Title: Evaluation of the Neonatal Autonomic Stress During Intubations Under Propofol in a Population of Premature Infants Under 33 w'GA
Acronym: PROPOSURF
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 18CH129; 2018-003233-14 (EudraCT Number)
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Hyaline Membrane Disease; Preterm Infant
Keywords: INSURE (Intubation / surfactant / extubation); LISA (Less-invasive surfactant administration); surfactant; propofol
MeSH Terms: conditions — Hyaline Membrane Disease; Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm neonates (< 33 weeks GA): Preterm neonates requiring in the first week of life, an elective tracheal intubation for surfactant administration by INSURE or LISA methods.
  Interventions: Other: electrocardiogram

INTERVENTIONS:
Other: electrocardiogram — Autonomic and hemodynamic evaluation with different indices (LF, heart rate, Systolic, diastolic and mean arterial blood pressure, SaO2) during a sedation protocol for intubation and surfactant administration according the INSURE or LISA technique.

SUMMARY:
Hyaline membrane disease is one of the leading causes of morbidity and mortality in premature newborns in industrialized countries. For 30 years, the management of the hyaline membranes disease has been transformed by intratracheal administration of exogenous surfactant (Curosurf®) at birth or in the following hours. In order to limit the harmful effects in terms of barotrauma of mechanical ventilation, several methods have been developed over the last decades, aiming at limiting the mechanical ventilation to the profile of non-invasive ventilation: Thus the administration of surfactant has become faster (although invasive) and if possible followed by immediate extubation following the INSURE (INtubation / SURfactant / Extubation) or LISA (Less-Invasive Surfactant Administration) procedure.

Given the fragility of the children concerned and their low weight, this invasive gesture has long been carried out without premedication. However, taking into account the pain induced and potential hemodynamic consequences of the gesture, neonatal societies now recommend the use of anesthetic before intubation, with a short duration sedative.

Propofol is a general anesthetic that combines these conditions and is widely used in pediatric anesthesia.

In that way, since 2016, the invetigators have modified the sedation protocol for intubation in our department and have recommended Propofol as first-line treatment for term and preterm newborn. A lot of study showed its hemodynamic safety in preterms. However, the investigators lack data on the autonomic stress really observed during intubation in this population. The investigators therefore propose to evaluate these physiological data in a non-randomized prospective observational study in premature infants under 33 weeks of gestational amenorrhea (GA), during a sedation protocol for intubation and surfactant administration according the INSURE or LISA technique, with standardized doses of propofol : 1mg/kg for preterm infants with a birthweight less than 1.5kg and 1.5mg/kg for higher birthweight.

ELIGIBILITY:
Inclusion Criteria:

* breathing rate > 60 cycles/min
* Silverman scale > 3 and < 6
* FiO2 > 30% and < 60%
* collected consent from parents

Exclusion Criteria:

* Preterm neonates with Intraventricular hemorrhage grade III & IV
* Preterm neonates with hemodynamic instability
* Preterm neonates with congenital heart disease
* Preterm neonates with severe congenital malformation
* Preterm neonates already sedated and/or under invasive mechanical ventilation
* FiO2 > 60%
* Silverman scale > 6
* Use of amines for maintaining blood pressure
* Use of sedatives or analgesics during the last 24 hours (except paracetamol and ibuprofen)

Max Age: 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm neonates (< 33 weeks GA) admitted to the tertiary Neonatal Intensive Care Unit of Saint-Etienne hospital requiring in the first week of life, an elective tracheal intubation for surfactant administration by INSURE or LISA methods
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Real-time LF values (low frequency) | during surfactant administration procedure
  * represent the well-being sympathetic activity of the autonomic nervous system
  * measured with electrocardiogram

SECONDARY OUTCOMES:
heart rate | during surfactant administration procedure
  - measured with electrocardiogram
systolic arterial blood pressure | during surfactant administration procedure
  - measured with a blood pressure cuff
diastolic arterial blood pressure | during surfactant administration procedure
  - measured with a blood pressure cuff
Oxygen saturation | during surfactant administration procedure
  - measured by pulse oximetry

CONTACTS AND LOCATIONS:
Overall Officials: Hugues PATURAL, Principal Investigator — CHU de Saint Etienne
Locations (1):
- CHU de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No